CLINICAL TRIAL: NCT00991653
Title: Weight Fluctuation After Breast Cancer Treatment
Status: Completed | Type: Observational
Sponsor: The Royal Bournemouth Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 08/H0201/35
Record Dates: First submitted 2009-10-06; First posted 2009-10-08 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer; Weight Gain
Keywords: Weight; Breast; Cancer
MeSH Terms: conditions — Breast Neoplasms; Weight Gain; Body Weight; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fasting blood sample to determine participants genotype, insulin and glucose levels.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Breast cancer: Diagnosed with breast cancer 1/1/2003 - 31/12/2007.
  Interventions: Procedure: Fasting blood sample.

INTERVENTIONS:
Procedure: Fasting blood sample. — Fasting blood sample taken following informed consent for genotyping, glucose and insulin levels.

SUMMARY:
This study aims to identify and quantify the factors associated with excess weight gain following treatment for breast cancer. It is believed that breast cancer patients gain more than 4% of their weight at diagnosis which is likely accompanied by an increase in body fat and waist circumference. It is further thought that this excess weight and increase in body fat and waist circumference are associated to tumour characteristics, chemotherapy, menopause status at diagnosis and the presence of genes related to obesity. It is also thought that women treated with chemotherapy have higher levels of glucose and insulin.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years of age or older.
* Diagnosed with breast cancer between 1/1/2003 and 31/12/2007.
* Able to understand and willing to sign informed consent.

Exclusion Criteria:

* Known diagnosis of previous breast/other cancer (other than completely resected non-melanoma skin cancer or successfully treated in situ cancer of the cervix.
* Known diagnosis of inflammatory bowel disease or malabsorption syndrome.
* Known diagnosis of endocrine problems associated with the development of obesity (cushings syndrome, hypo/hyperthyroid, thyroiditis)
* Treatment for psychiatric disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females over 18 years diagnosed with breast cancer between 1/1/2003 and 31/12/2007.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2008-08; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To provide evidence of the relationship between weight gain following diagnosis of breast cancer and tumour characteristics, chemotherapy, menopause status at diagnosis and the presence of genes related to obesity. | 12-18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Tamas Hickish, Principal Investigator — Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust